CLINICAL TRIAL: NCT01276470
Title: Environmental Risk Factors for the Anti-Synthetase Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110072; 11-E-0072
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-04-14

CONDITIONS: Myositis; Dermatomyositis; Polymyositis; Juvenile Dermatomyositis; Juvenile Polymyositis
Keywords: Adult and Pediatric Autoimmune Disease; Antibody; Autoimmune Diseases; Autoimmunity Pathogenesis; Environmental Risk Factors; Natural History
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Antisynthetase Negative: Subjects with myositis without antisynthetase syndrome
- Antisynthetase Positive: Subject with myositis with antisynthetase syndrome
- Healthy Control: Subjects without autoimmune disease

SUMMARY:
Background:

* Like other complex diseases, autoimmune diseases are the result of numerous causes, including genetic and environmental factors. Some researchers believe that people who are susceptible to autoimmune disorders develop them when the body reacts to environmental or other factors by creating white blood cells that attack the body s own tissues, which then progresses to autoimmune diseases. These immune-triggered disorders can overlap with one another to some extent, but most autoimmune diseases have certain distinct triggers.
* The autoimmune disorder myositis weakens the muscles and may cause other health problems. Environmental exposures associated with myositis include ultraviolet radiation, stressful life events and muscle overexertion, collagen implants, infections such as retroviruses and streptococci bacteria, and certain drugs and chemicals. Some individuals with myositis also produce proteins in the blood called autoantibodies that react with certain parts of the person s own cells, called synthetases, which are involved in making new proteins. A syndrome called the anti-synthetase syndrome, which includes myositis and lung disease, is associated with having the anti-synthetase autoantibodies. Researchers are interested in studying differences in environmental exposures in individuals with myositis. This study is being conducted to determine if persons with the anti-synthetase syndrome have had different environmental exposures before disease onset compared with other patients with myositis who do not have this syndrome and also compared with healthy volunteers.

Objectives:

- To determine whether selected infectious and noninfectious environmental exposures are more common in individuals who have myositis with the anti-synthetase syndrome, compared with healthy volunteers.

Eligibility:

- Individuals who have been diagnosed with myositis (with or without anti-synthetase autoantibodies), and healthy volunteers without autoimmune disorders.

Design:

* Participants will be screened with a full medical history and physical examination, and will provide blood, urine and house dust samples.
* Participants will complete questionnaires about their medical history and the types of exposures they have had at work, at home, and elsewhere. Participants who have myositis will also be asked about certain infections, heavy exercise or physical exertion, sun exposure, tobacco and alcohol use, and stressful events prior to being diagnosed with the disease. Healthy volunteers will be asked about the same exposures before the date of diagnosis of disease of the myositis subject to which they have been matched.
* Participants will receive a kit that contains instructions and a filter to be put onto their vacuum cleaner to collect house dust in the bedroom. This dust will be kept for possible future analyses of infectious or toxic agents based on the other results from the study.
* Individuals with myositis will have other tests as clinically indicated, including lung function tests and imaging studies.

DETAILED DESCRIPTION:
Most autoimmune diseases are thought to develop as a result of chronic immune activation and dysregulation after selected environmental exposures in genetically susceptible individuals. Based on prior studies suggesting roles for noninfectious and infectious agents in the development of myositis, as well as the known clinical, epidemiologic and genetic differences among phenotypes, we hypothesize that different myositis phenotypes are triggered by different environmental exposures in genetically susceptible individuals. One phenotype that is particularly well-defined clinically and genetically, and for which environmental triggers are likely, is myositis associated with anti-synthetase autoantibodies (defined as the anti-synthetase syndrome). These patients have an acute myositis onset in the spring of the year and also tend to develop fevers, elevated white blood cell counts, arthritis and interstitial lung disease. Although these features are consistent with an environmental trigger for the anti-synthetase syndrome, and although case reports and animal models suggest infectious or noninfectious agents may play a role, no study has systematically assessed environmental agents in this population.

In collaboration with multiple centers, we plan to test the hypothesis that certain environmental exposures are associated with the anti-synthetase syndrome and differ from those seen in matched controls and in myositis patients without the anti-synthetase syndrome. The specific aims of this study are to: 1) determine whether selected noninfectious environmental exposures are more common preceding disease onset in 150 recent-onset (defined as within 24 months of meeting criteria for possible, probable or definite myositis) myositis patients with the anti-synthetase syndrome, compared with 150 control subjects without autoimmune disease (1:1 matched with the patients), and compared with 150 recent-onset myositis patients without the anti-synthetase syndrome; and 2) determine whether selected infectious agents can be detected more frequently in blood samples of recent-onset anti-synthetase syndrome patients compared with matched controls, and in blood or biopsy samples from recent-onset anti-synthetase myositis patients compared with recent-onset myositis patients without the anti-synthetase syndrome.

Medical histories, concurrent conditions and environmental questionnaire information will be collected from all participants. Subjects will undergo a clinical, laboratory and immunologic assessment to document current diagnoses, disease manifestations and severity. A chest x-ray, high resolution computed tomography (HRCT) of the chest, pulmonary function tests, bronchoalveolar lavage, and muscle and lung biopsies will be performed as clinically indicated. Blood DNA and RNA sera, biopsy and house dust repositories will be created for current and future investigations.

ELIGIBILITY:
* INCLUSION CRITERIA:

There are no gender or ethnic restrictions to enrollment in the study. Age restrictions for children do apply to enrollment in the study.

The inclusion criteria for enrollment of myositis subjects are:

1. Diagnosis of myositis based on criteria for possible, probable or definite PM or DM, with or without other connective tissue diseases, documented within 24 months of enrollment (using the most recent diagnosis date to define the 24-month period).
2. CXR to assess possible ILD and assign the subject to the presumptive anti-synthetase positive or negative category if clinically indicated.
3. Children must be greater than two years of age.
4. Able and willing to give informed consent, to complete the questionnaires and to donate blood samples (in case of children greater than 2 years of age but <18 years of age, parent/legal guardian must be willing and able to provide informed consent and child will provide assent according to child s maturity level and understanding).

The exclusion criteria for myositis subjects are:

1. Cancer-associated myositis (cancer diagnosed within 2 years of the diagnosis of myositis).
2. Inclusion body myositis.
3. Myositis that has clearly developed as the result of a drug, toxin or other exposure and has resolved after discontinuation of the exposure to that agent.
4. Children less than 2 years of age.

The inclusion criteria for controls are:

1. Friends or, if friends are not available, cousins of the anti-synthetase-positive myositis patient, or, if friends or cousins are not available, volunteers from the general community (such as the NIH Normal volunteer program), race- gender- and age- (within 5 years for minors and within 10 years for adults) matched, and when possible who is living as close as possible to the geographic area of the myositis patient.
2. Controls should be without a recognized autoimmune disease or ILD.
3. Able and willing to give informed consent, to complete the questionnaires and to donate blood samples (in case of children greater than 2 years of age but <18 years of age, parent/legal guardian must be willing and able to provide informed consent) and child will provide assent according to child maturity level and understanding).

The exclusion criteria for all protocol subjects are:

1. Medical illness that in the judgment of the investigators does not allow safe blood draws or other clinical evaluations needed for study participation.
2. Cognitive impairment.
3. Not able or willing to give informed assent or consent.
4. Children less than 2 years of age.
5. Patients who at their reference date were not in the US or Canada
6. Individuals currently incarcerated

HIV considerations:

HIV is not an exclusion for affected participants in this study for the two following reasons:

1. It has no impact on study procedures or tests.
2. It may be one of the viral risk factors we are investigating.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population; There are no gender or ethnic restrictions to enrollment in the study. Age restrictions for children do apply to enrollment in the study.@@@@@@
Sampling Method: Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2011-02-09 (Actual)

PRIMARY OUTCOMES:
To determine whether selected noninfectious environmental exposures are more common prior to disease in recent-onset pts. w/anti-sythetase syndrome compared w/controls w/o autoimmune disease (1:1 matched with the pts.) and compared w/recent-onse... | Enrollment
  Environmental Questionnaire (EQ) and Child Environmental Questionnaire (CQ)

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Schiffenbauer, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (8):
- United States (8):
  - University of Miami Hospital, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Mid-Atlantic Kaiser Permanente, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-E-0072.html